CLINICAL TRIAL: NCT00668447
Title: Soy Proteins and Isoflavones Impact Bone Mineral Density in Older Women
Brief Title: Soy and Isoflavones Effect on Bone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: University of Connecticut (Other)
Responsible Party: Anne Kenny, MD, Associate Professor of Medicine, University of Connecticut Center on Aging
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0102; USDA CONR-2001-00630
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Osteoporosis
Keywords: bone density; bone loss; postmenopausal
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Soy protein and isoflavone tablets
  Interventions: Dietary Supplement: Soy Isolate; Dietary Supplement: Novasoy isoflavones
- 2 (Active Comparator): Soy protein and placebo tablets
  Interventions: Dietary Supplement: Soy Isolate; Dietary Supplement: Placebo tablets
- 3 (Active Comparator): control protein and Isoflavone tablets
  Interventions: Dietary Supplement: Control protein; Dietary Supplement: Novasoy isoflavones
- 4 (Placebo Comparator): control protein and placebo tablets
  Interventions: Dietary Supplement: Control protein; Dietary Supplement: Placebo tablets

INTERVENTIONS:
Dietary Supplement: Soy Isolate — 20 grams of powder mixed in beverages or food daily for one year
  Other Names: Pro Fam 930, 066-930
  Arms: 1; 2
Dietary Supplement: Control protein — 20 grams of powder mixed in beverages or food daily for one year
  Arms: 3; 4
Dietary Supplement: Novasoy isoflavones — 3 tablets daily for one year
  Arms: 1; 3
Dietary Supplement: Placebo tablets — 3 tablets daily for one year
  Arms: 2; 4

SUMMARY:
The purpose of this study is to test the effect of 1 year of added dietary soy protein and/or soy isoflavones on bone mineral density in late postmenopausal women.

DETAILED DESCRIPTION:
Although soy foods contain several components (isoflavones and amino acids) that could potentially have positive effects on bone health, there are few long term, large, clinical trials using soy as a means of improving bone mineral density. The objective of this study is to provide daily soy protein and isoflavones to healthy older women in order to answer three major questions:

1. Does soy protein alone affect bone metabolism?
2. Do isoflavones, given with soy protein, affect bone metabolism?
3. What dose of isoflavones affects bone in older women?

We hypothesize that soy protein will have a beneficial effect on bone in older women compared to control protein. Further, we hypothesize that there will be an additional benefit to bone in women who receive soy protein plus isoflavones (at both doses) compared to soy protein alone.

Both control and soy proteins used in the study were isolates, meaning they were the highest concentration of protein (85-90% by weight) in order to minimize the volume of protein supplement that each woman was asked to ingest on a daily basis. The soy protein was an alcohol-washed, soy protein isolate containing 90% protein and negligible isoflavone (0.2 mg/g product). The control protein was a mix consisting of 50% protein from sodium caseinate, 25% protein from whey protein and 25% from egg white protein. The use of a mix of proteins as a control provides a more balanced level of amino acids, mimics the real life mix of proteins that humans typically consume, and avoids the unique characteristics of one source of protein. In order to maintain the dietary protein intake constant, the participant was counseled to decrease her intake of other sources of protein from primarily animal sources by approximately 3 ounces per day (the approximate equivalent of the protein powders). The isoflavones tablets each contained 57 mg of total isoflavone from primarily genistein, glycitein, and daidzein and their beta-glycosides.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women 65 years old or older
* Able to travel to the clinical sites for follow-up visits

Exclusion Criteria:

* History of disease that may affect bone metabolism (including Paget's disease, primary hyperparathyroidism, osteomalacia, untreated hyperthyroidism, or multiple myeloma)
* Cancer of any kind (except basal or squamous cell of skin) in past 5 years
* Use of any of the following medications within the past 2 years: calcitonin, calcitriol, heparin, phenytoin, phenobarbital
* Use at any time of bisphosphonates, long-term corticosteroids (over 6 months), methotrexate, or fluoride
* Estimated creatinine clearance less than 50 ml/min
* History of chronic liver disease or evidence of liver disease on screening
* History of hip fracture
* Known vertebral fracture within the past year
* Vegans

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2001-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Bone turnover markers | baseline, 3 months, and 1 year

SECONDARY OUTCOMES:
Bone Mineral Density | Baseline, 6 and 12 months
Quality of life measured by Medical Outcomes Short Form | Baseline, 6 and 12 months
Medication Side Effects | 3 , 6, 9, and 12 months
Adherence to dietary intervention through the use of 24-hour recall | 3, 6, 9, and 12 months
Long-term medication behavior self-efficacy scale | 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kerstetter, PhD, Principal Investigator — Department of Allied Health Sciences, University of Connecticut
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Evans EM, Racette SB, Van Pelt RE, Peterson LR, Villareal DT. Effects of soy protein isolate and moderate exercise on bone turnover and bone mineral density in postmenopausal women. Menopause. 2007 May-Jun;14(3 Pt 1):481-8. doi: 10.1097/01.gme.0000243570.78570.f7. PMID 17213752
- [Background] Alekel DL, Germain AS, Peterson CT, Hanson KB, Stewart JW, Toda T. Isoflavone-rich soy protein isolate attenuates bone loss in the lumbar spine of perimenopausal women. Am J Clin Nutr. 2000 Sep;72(3):844-52. doi: 10.1093/ajcn/72.3.844. PMID 10966908
- [Background] Arjmandi BH, Lucas EA, Khalil DA, Devareddy L, Smith BJ, McDonald J, Arquitt AB, Payton ME, Mason C. One year soy protein supplementation has positive effects on bone formation markers but not bone density in postmenopausal women. Nutr J. 2005 Feb 23;4:8. doi: 10.1186/1475-2891-4-8. PMID 15727682
- [Derived] Kenny AM, Mangano KM, Abourizk RH, Bruno RS, Anamani DE, Kleppinger A, Walsh SJ, Prestwood KM, Kerstetter JE. Soy proteins and isoflavones affect bone mineral density in older women: a randomized controlled trial. Am J Clin Nutr. 2009 Jul;90(1):234-42. doi: 10.3945/ajcn.2009.27600. Epub 2009 May 27. PMID 19474141